CLINICAL TRIAL: NCT02396550
Title: Influence of Patient Expectations With Lateral Epicondylalgia in Applying Mobilization With Movement. Clinical Trial
Brief Title: Influence of Patient Expectations With Lateral Epicondylalgia in Applying Mobilization With Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Raúl Ferrer Peña, Prof., Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PI-1900
Record Dates: First submitted 2015-03-11; First posted 2015-03-24 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Tennis Elbow
Keywords: Expectations
MeSH Terms: conditions — Tennis Elbow | interventions — Movement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Positive Expectations (Experimental): Procedure/Surgery: Mobilization with movement in patients with lateral epicondylalgia with modification of its expectations into positive
  Interventions: Behavioral: Positive Expectations; Procedure: Mobilization with movement
- Neutral Expectations (Experimental): Procedure/Surgery: Mobilization with movement in patients with lateral epicondylalgia with modification of its expectations into neutral
  Interventions: Procedure: Mobilization with movement

INTERVENTIONS:
Behavioral: Positive Expectations — Give positive expectation of the treatment efficacy to patients
  Arms: Positive Expectations
Procedure: Mobilization with movement — Give neutral expectation of the treatment efficacy to patients

SUMMARY:
Lateral epicondylalgia affects people of both gender between 1 and 3% of the world population, with up to 15% in the working population reaching an average of 12 weeks off work for this reason. One of the conservative treatments that have shown effective is the mobilization with movement, whose mechanisms of action are not known. According Bialosky et al., possible effects of manual therapy are based on the neurophysiological mechanisms at peripheral, spinal and supraspinal level. Among the mechanisms to supraspinal level is the placebo effect, which is influenced by psychological factors such as conditioning and expectations.

Changing expectations to determine the influence on the treatment has been studied in healthy subjects, showing improvement with positive expectations and worsening to negative and neutral expectations.

However the result of modifying the previous expectations for treatment in patients with pain has not been studied.

The aim of our study is to test the influence that positive expectations have on the effectiveness of treatment with mobilization with movement in patients with lateral epicondylalgia.

ELIGIBILITY:
Inclusion Criteria:

* Lateral Epicondylalgia Diagnosis

Exclusion Criteria:

* Previous Treatment with Manual Therapy
* Previous Treatment with injection 6 months before
* Radiculopathy
* Bilateral Symptoms
* Fracture

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 0 - 10 days
  measured with the Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Threshold Pressure Pain | 0 - 10 days
  measured with algometry
Perceived Disability | 0-10 days
  with the DISABILITIES OF THE ARM, SHOULDER AND HAND (DASH) Questionnaire
Kinesiophobia | 0 - 10 days
  with the Tampa Scale of Kinesiophobia

CONTACTS AND LOCATIONS:
Locations (1):
- Raúl Ferrer Peña, Arganda, Madrid, Spain

REFERENCES:
- [Background] Bialosky JE, Bishop MD, George SZ, Robinson ME. Placebo response to manual therapy: something out of nothing? J Man Manip Ther. 2011 Feb;19(1):11-9. doi: 10.1179/2042618610Y.0000000001. PMID 22294849
- [Background] Bialosky JE, Bishop MD, Robinson ME, Barabas JA, George SZ. The influence of expectation on spinal manipulation induced hypoalgesia: an experimental study in normal subjects. BMC Musculoskelet Disord. 2008 Feb 11;9:19. doi: 10.1186/1471-2474-9-19. PMID 18267029
- [Background] Bialosky JE, George SZ, Horn ME, Price DD, Staud R, Robinson ME. Spinal manipulative therapy-specific changes in pain sensitivity in individuals with low back pain (NCT01168999). J Pain. 2014 Feb;15(2):136-48. doi: 10.1016/j.jpain.2013.10.005. Epub 2013 Oct 27. PMID 24361109
- [Background] Paungmali A, O'Leary S, Souvlis T, Vicenzino B. Hypoalgesic and sympathoexcitatory effects of mobilization with movement for lateral epicondylalgia. Phys Ther. 2003 Apr;83(4):374-83. PMID 12665408
- [Background] Vicenzino B, Paungmali A, Buratowski S, Wright A. Specific manipulative therapy treatment for chronic lateral epicondylalgia produces uniquely characteristic hypoalgesia. Man Ther. 2001 Nov;6(4):205-12. doi: 10.1054/math.2001.0411. PMID 11673930